CLINICAL TRIAL: NCT06814093
Title: Robotic Versus Laparoscopic Surgery for Middle and Low Rectal Cancer: A Retrospective Cohort Study Emulating the Target Trial
Brief Title: Robotic Versus Laparoscopic Surgery for Middle and Low Rectal Cancer: a Target Trial Emulation
Status: Active, not recruiting | Type: Observational
Sponsor: Xu jianmin (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Director of Colorectal Surgery, Fudan University
Organization: Fudan University (Other)
Other Study IDs: CCS-DASET-TTE-REAL
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Robotic Surgical Procedures; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic group: Patients received robotic surgery for middle and low rectal cancer
  Interventions: Procedure: Robotic surgery
- Laparoscopic group: Patients received laparoscopic surgery for middle and low rectal cancer
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Robotic surgery — Robotic surgery for radical resection of middle and low rectal cancer
  Groups: Robotic group
Procedure: Laparoscopic surgery — Laparoscopic surgery for radical resection of middle and low rectal cancer
  Groups: Laparoscopic group

SUMMARY:
This study aims to compare the effectiveness of robotic surgery versus laparoscopic surgery in treating low rectal cancer. While robotic surgery has gained popularity, there is limited long-term evidence regarding its outcomes. By using real-world data from a specialized multicenter colorectal cancer database in Shanghai, China, this retrospective cohort study will emulate the target trial to evaluate whether robotic surgery offers advantages over laparoscopic surgery. Key factors such as disease-free survival, locoregional recurrence, circumferential margin positivity, and postoperative complications will be examined. The goal is to provide stronger, evidence-based support for the clinical use of robotic surgery in treating low rectal cancer.

ELIGIBILITY:
Inclusion criteria:

1. Age from 18 years to 80 years;
2. American Society of Anesthesiologists (ASA) class I - III;
3. Histologically proved rectal adenocarcinoma;
4. Inferior tumor edge ≤ 10 cm from anal verge, measured by rigid rectoscopy;
5. Tumor assessed as cT1-T3 (mesorectal fascia not involved) N0-1, or ycT1-T3 Nx after preoperative radio- or chemoradiotherapy, measured by pelvic MRI;
6. No evidence of distant metastases (including pelvis, peritoneum, liver, lung, brain, bone, distant lymph node, etc), according to ultrasound, CT, MRI, PET-CT, etc;
7. No other malignancies in medical history except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri;
8. Received either robotic or laparoscopic surgery; 9） Surgery with radical intent;

10) Informed consent.

Exclusion criteria

1. Emergency surgery for acute intestinal obstruction, bleeding, perforation, etc;
2. Synchronous colon surgery for multiple colorectal tumors or other schedules;
3. Hereditary colorectal cancer (familial adenomatosis polyposis, Lynch Syndrome, etc.);
4. Co-existent inflammatory bowel disease;
5. Pregnancy or lactation;
6. Patients received treatment other than preoperative radio- or chemoradiotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data is sourced from the Colorectal Cancer Specialty Cohort Database and Biobank, established through the "Construction and Application of the Shanghai Colorectal Cancer Specialty Cohort Database and Biobank" project. The research will utilize cohort data collected from January 2021 to May 2022 (17 months). This specialized database was led by Zhongshan Hospital, Fudan University, in collaboration with Shanghai Tenth People's Hospital, Fudan University Shanghai Cancer Center, First Affiliated Hospital of Naval Medical University (Changhai Hospital), Renji Hospital, Shanghai Jiao Tong University School of Medicine, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, and Shanghai First People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2702 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
3-year postoperative disease-free survival rate | From surgery to three years postoperatively
  Disease-free survival event is defined as any death or locoregional recurrence or distant metastases.

SECONDARY OUTCOMES:
Circumferential resection margin positivity rate | 14 days during postoperative pathological examination
  Circumferential resection margin positivity is defined as 1 mm or less from the tumor.
30-day postoperative complication rate (Clavien-Dindo grade 2 or higher grade) | From surgery to 30 days postoperatively
  30-day postoperative complication rate is defined according to the Clavien-Dindo grade system. Only complications in grade 2 or higher grade will be calculated.
rate of abdominoperineal resection | 30 days after surgery
  percentage of patients received abdominoperineal resection
3-year postoperative locoregional recurrence rate | From surgery to three years postoperatively
  Locoregional recurrence is defined as any cancer recurrence in the pelvic or perineal area.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No